CLINICAL TRIAL: NCT02796391
Title: Facilitating Smoking Cessation With Reduced Nicotine Cigarettes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: James and Esther King Biomedical Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MCC-18671
Record Dates: First submitted 2016-06-03; First posted 2016-06-10 (Estimated); Results first posted 2022-10-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Smoking Cessation
Keywords: nicotine; cigarettes; very low nicotine content (VLNC); smoking cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Products

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Study 1: Immediate Reduction (Experimental): Participants will receive cigarettes with the lowest nicotine dose (.03 mb nicotine yield). They will receive a targeted intervention workbook ("Count down: Preparing to Quit Smoking with Low-Nicotine Cigarettes") and will be provided with one-on-one counseling.
  Interventions: Drug: Very Low Nicotine Content (VLNC) Cigarettes; Behavioral: One on One Counseling
- Study 1: Gradual Reduction (Experimental): Participants will receive VLNC (very low nicotine cigarettes) containing nicotine yields of .7 mg for week 1, .26 mg for week 2, .12 for week 3, and .03 for week 4.They will receive a targeted intervention workbook ("Count down: Preparing to Quit Smoking with Low-Nicotine Cigarettes") and will be provided with one-on-one counseling.
  Interventions: Drug: Very Low Nicotine Content (VLNC) Cigarettes; Behavioral: One on One Counseling
- Study 2: Targeted/Immediate Reduction (Experimental): Participants will receive VLNC (very low nicotine cigarettes) containing nicotine yields of .7 mg for week 1, .26 mg for week 2, .12 for week 3, and .03 for week 4.They will receive a targeted intervention workbook ("Count down: Preparing to Quit Smoking with Low-Nicotine Cigarettes") and will be provided with one-on-one counseling.
  Interventions: Drug: Very Low Nicotine Content (VLNC) Cigarettes; Behavioral: One on One Counseling
- Study 2: Targeted/Gradual Reduction (Experimental): Participants will receive VLNC (very low nicotine cigarettes) containing nicotine yields of .7 mg for week 1, .26 mg for week 2, .12 for week 3, and .03 for week 4. Participants will also receive targeted materials (booklet series entitled ("Count down: Preparing to Quit Smoking with low-Nicotine Cigarettes") as well as one-on-one counseling.
  Interventions: Drug: Very Low Nicotine Content (VLNC) Cigarettes; Behavioral: One on One Counseling
- Study 2: Generic/Immediate Reduction (Experimental): Participants will receive VLNC (very low nicotine cigarettes) with the lowest nicotine dose (.03 mb nicotine yield). Participants will also receive the generic ("Clearing the Air") materials, as well as one-on-one counseling.
  Interventions: Drug: Very Low Nicotine Content (VLNC) Cigarettes; Behavioral: One on One Counseling
- Study 2: Generic/Gradual Reduction (Experimental): Participants will receive VLNC (very low nicotine cigarettes) containing nicotine yields of .7 mg for week 1, .26 mg for week 2, .12 for week 3, and .03 for week 4. Participants will also receive the generic ("Clearing the Air") materials, as well as one-on-one counseling.
  Interventions: Drug: Very Low Nicotine Content (VLNC) Cigarettes; Behavioral: One on One Counseling

INTERVENTIONS:
Drug: Very Low Nicotine Content (VLNC) Cigarettes — Eligible participants will receive a 1-week supply (based on typical # cigarettes/day x 1.5) of normal nicotine content (NNC) (.8 mg nicotine yield) study cigarettes to smoke exclusively during one baseline week.
  Study 1: Participants (n=20) will then be randomly selected to receive either the lowest nicotine dose of VLNC cigarettes, or gradual decreasing nicotine VLNC cigarettes, ten participants per each group, over the next four weeks.
  Study 2: Participants (n=208) will be randomly assigned to 1 of 4 Study 2 Reduction Arms, 52 participants per arm.
  Other Names: SPECTRUM®; Research Cigarettes; NOT-DA-13-002
Behavioral: One on One Counseling — All participants will receive One on One Counseling.

SUMMARY:
STUDY 1: INTERVENTION DEVELOPMENT The purpose of this study is to determine the best way to help people stop smoking by using very low nicotine content (VLNC) cigarettes. This developmental pilot study (n=20) will determine the feasibility of the treatment approach and methodology using a targeted intervention, and lead to refinements for a subsequent randomized controlled trial (RCT).

STUDY 2: RANDOMIZED CONTROLLED TRIAL The purpose of this study is to see if a targeted intervention will help people to stop or reduce smoking better than a standard intervention using very low nicotine content (VLNC) cigarettes, and to determine the optimal nicotine tapering schedule (gradual vs. immediate) during a 5-week pre-quit period. About 208 participants will take part in this phase of the study at Moffitt Cancer Center.

DETAILED DESCRIPTION:
The current project will (1) develop a theory-based, user-friendly, and efficient set of targeted cessation materials to facilitate extinction during pre-quit VLNC smoking, (2) establish the feasibility of recruitment and measurement strategies to be used in the RCT, (3) determine whether immediate vs. gradual pre-quit nicotine tapering in combination with the targeted behavioral intervention has beneficial effects (on cessation-related and intermediate outcomes) for eventual comparison with validated cessation methods (e.g., NRT), and (4) examine several potential moderators and mediators of treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* smoke at least 5 cigarettes daily for the past year
* expired-air carbon monoxide (CO) > 8 ppm (if ≤ 8 ppm, then NicAlert Strip > 2)
* current motivation to quit smoking
* able to speak and read English sufficiently for completion of consent form and questionnaires
* 18 years of age or older

Exclusion Criteria:

* pregnant or breastfeeding
* significant unstable medical/psychiatric or substance use disorders, or medically/psychiatrically at risk in the judgment of the study physician or principal investigator (PI)
* positive urine screen for cocaine, opiates, methadone, benzodiazepines, barbiturates, amphetamines, methamphetamines, or PCP (NOTES: THC will be tested but will not be an exclusionary criterion; participants with valid prescriptions for opiates, benzodiazepines, barbiturates, amphetamines or methadone will not be excluded; participants failing the toxicology screen will be allowed to re-screen once)
* breath alcohol level > 0.01 (one re-screen allowed)
* binge alcohol drinking (4/5 [female/male] drinks per day more than 9 days in the past month)
* systolic/diastolic blood pressure (BP) greater than or equal to 160/100, or below 90/50 (one re-screen allowed)
* heart rate greater than or equal to 105 beats per minute (bpm), or below 45 bpm (one re-screen allowed)
* ever used reduced nicotine cigarettes
* smoke 'roll your own' cigarettes exclusively
* used smoking cessation medications within the past three months
* are currently enrolled in a smoking cessation program
* actively trying to quit
* used other tobacco products (including e-cigarettes more than 9 days in the past month
* currently taking the following medications: Phenytoin [Brand Name: Dilantin]; Carbamazepine [Brand Name: Tegretol, Carbatrol, Equetro, Epitol]; Oxcarbazepine [Brand Name: Trileptal]; Primidone [Brand Name: Mysoline]; Phenobarbital; Bendamustine (Treanda); Clopidogrel (Plavix); Clozapine (Clozaril, FazaClo); Erlotinib (Tarceva); Flecainide (Tambocor); Fluvoxamine (Luvox); Irinotecan (Camptosar); Olanzapine (Zyprexa); Ropinirole (Requip); Tacrine (Cognex); Theophylline (Theo Dur, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vani Simmons, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant did not meet inclusion criteria in study 1 before being assigned to an arm.
Groups:
- Study 1: Gradual Reduction: Participants will receive very low nicotine cigarettes containing nicotine yields of .7 mg for week 1, .26 mg for week 2, .12 for week 3, and .03 for week 4.They will receive a targeted intervention workbook ("Count down: Preparing to Quit Smoking with Low-Nicotine Cigarettes") and will be provided with one-on-one counseling.
- Study 2: Targeted/Immediate Reduction: Participants will receive cigarettes with the lowest nicotine dose (.03 mb nicotine yield). Participants will also receive targeted materials (booklet series entitled ("Count down: Preparing to Quit Smoking with low-Nicotine Cigarettes") as well as one-on-one counselling.
- Study 2: Targeted/Gradual Reduction: Participants will receive very low nicotine cigarettes containing nicotine yields of .7 mg for week 1, .26 mg for week 2, .12 for week 3, and .03 for week 4. Participants will also receive targeted materials (booklet series entitled ("Count down: Preparing to Quit Smoking with low-Nicotine Cigarettes") as well as one-on-one counseling.
- Study 2: Generic/Immediate Reduction: Participants will receive cigarettes with the lowest nicotine dose (.03 mb nicotine yield). Participants will also receive the generic ("Clearing the Air") materials, as well as one-on-one counseling.
- Study 2: Generic/Gradual Reduction: Participants will receive very low nicotine cigarettes containing nicotine yields of .7 mg for week 1, .26 mg for week 2, .12 for week 3, and .03 for week 4. Participants will also receive the generic ("Clearing the Air") materials, as well as one-on-one counseling.
Period: Overall Study
Arm/Group | Study 1: Immediate Reduction | Study 1: Gradual Reduction | Study 2: Targeted/Immediate Reduction | Study 2: Targeted/Gradual Reduction | Study 2: Generic/Immediate Reduction | Study 2: Generic/Gradual Reduction
Started | 7 | 8 | 41 | 32 | 34 | 40
Completed | 4 | 5 | 16 | 14 | 14 | 20
Not Completed | 3 | 3 | 25 | 18 | 20 | 20
Not completed — Lost to Follow-up | 2 | 2 | 13 | 8 | 14 | 13
Not completed — COVID | 0 | 0 | 5 | 5 | 2 | 4
Not completed — Participant did not like study cigarettes | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 4 | 3 | 4 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study 1: Immediate Reduction | Study 1: Gradual Reduction | Study 2: Targeted/Immediate Reduction | Study 2: Targeted/Gradual Reduction | Study 2: Generic/Immediate Reduction | Study 2: Generic/Gradual Reduction | Total
Number analyzed (Participants) | 7 | 8 | 41 | 32 | 34 | 40 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 8 | 31 | 29 | 30 | 34 | 137
  >=65 years | 2 | 0 | 10 | 3 | 4 | 6 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 23 | 20 | 19 | 22 | 90
  Male | 4 | 5 | 18 | 12 | 15 | 18 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 5 | 6 | 3 | 5 | 20
  Not Hispanic or Latino | 7 | 7 | 36 | 26 | 31 | 35 | 142
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 4 | 2 | 4 | 4 | 17
  White | 5 | 6 | 35 | 28 | 28 | 34 | 136
  More than one race | 0 | 0 | 1 | 2 | 0 | 1 | 4
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 41 | 32 | 34 | 40 | 162

OUTCOME MEASURES:

1. Primary Outcome: Study 1 - Rate of Participant Completion of Pilot
Description: Pilot: Complete formative research based on 15 participants to prepare for Study 2.
Time Frame: Up to 2 Weeks
Measure: Count of Participants; unit: Participants
Groups:
- Study 1: Immediate Reduction: This group will receive the lowest nicotine dose (.03 mb nicotine yield) very low nicotine content (VLNC) cigarettes, each of four pre-quit weeks (immediate reduction.
  Study 1: Participants will be randomly assigned to 1 of 2 groups (Immediate or gradual nicotine reduction). They will all receive a targeted intervention workbook ("Countdown: Preparing to Quit Smoking with Low-Nicotine Cigarettes") and will be provided with brief one-on-one counseling.
  Very Low Nicotine Content (VLNC) Cigarettes: Eligible participants will receive a 1-week supply (based on typical # cigarettes/day x 1.5) of normal nicotine content (NNC) (.8 mg nicotine yield) study cigarettes to smoke exclusively during one baseline week.
  Study 1: Participants (n=20) will then be randomly selected to receive either the lowest nicotine dose of VLNC cigarettes, or gradual decreasing nicotine VLNC cigarettes, ten participants per each group, over the next four weeks.
  Study 2: Participants (n=208) will be randomly assigned to 1 of 4 Study 2 Reduction Arms, 52 participants per arm.
  One on One Counseling: All participants will receive One on One Counseling.
- Study 1: Gradual Reduction: This group will receive VLNC cigarettes containing nicotine yields of .7 mg for week 1, .26 mg for week 2, .12 for week 3, and .03 for week 4 (gradual reduction).
  Study 1: Participants will be randomly assigned to 1 of 2 groups (Immediate or gradual nicotine reduction). They will all receive a targeted intervention workbook ("Countdown: Preparing to Quit Smoking with Low-Nicotine Cigarettes") and will be provided with brief one-on-one counseling.
  Very Low Nicotine Content (VLNC) Cigarettes: Eligible participants will receive a 1-week supply (based on typical # cigarettes/day x 1.5) of normal nicotine content (NNC) (.8 mg nicotine yield) study cigarettes to smoke exclusively during one baseline week.
  Study 1: Participants (n=20) will then be randomly selected to receive either the lowest nicotine dose of VLNC cigarettes, or gradual decreasing nicotine VLNC cigarettes, ten participants per each group, over the next four weeks.
  Study 2: Participants (n=208) will be randomly assigned to 1 of 4 Study 2 Reduction Arms, 52 participants per arm.
  One on One Counseling: All participants will receive One on One Counseling.
Arm/Group | Study 1: Immediate Reduction | Study 1: Gradual Reduction
Number analyzed (Participants) | 7 | 8
Participants | 4 | 5

2. Primary Outcome: Study 2 - Participant Abstinence Success at 2 Months
Description: Participants reporting 7-day point prevalence abstinence at 2 months
  RCT: The purpose of Study 2 is to test effects of the targeted intervention developed in Study 1 on smoking cessation. Comparison of abstinence success per treatment arm, utilizing 7-day point prevalence abstinence at each follow-up assessment.
Time Frame: At 2 Months
Measure: Number; unit: participants
Groups:
- Study 2: Targeted/Immediate Reduction; Study 2: Generic/Immediate Reduction: This group will receive the lowest nicotine dose (.03 mg nicotine yield) very low nicotine content (VLNC) cigarettes, each of four pre-quit weeks (immediate reduction).
  Study 2: Participants will be randomly assigned to 1 of 4 groups (Immediate or gradual nicotine reduction/ Generic or targeted intervention). They will receive either targeted ("Countdown: Preparing to Quit Smoking with Low-Nicotine Cigarettes") or generic ("Clearing the Air") materials, and will receive one-on-one counseling.
  Very Low Nicotine Content (VLNC) Cigarettes: Eligible participants will receive a 1-week supply (based on typical # cigarettes/day x 1.5) of normal nicotine content (NNC) (.8 mg nicotine yield) study cigarettes to smoke exclusively during one baseline week.
  Study 1: Participants (n=20) will then be randomly selected to receive either the lowest nicotine dose of VLNC cigarettes, or gradual decreasing nicotine VLNC cigarettes, ten participants per each group, over the next four weeks.
  Study 2: Participants (n=208) will be randomly assigned to 1 of 4 Study 2 Reduction Arms, 52 participants per arm.
  One on One Counseling: All participants will receive One on One Counseling.
- Study 2: Targeted/Gradual Reduction; Study 2: Generic/Gradual Reduction: This group will receive VLNC cigarettes containing nicotine yields of .7 mg for week 1, .26 mg for week 2, .12 for week 3, and .03 for week 4 (gradual reduction).
  Study 2: Participants will be randomly assigned to 1 of 4 groups (Immediate or gradual nicotine reduction/ Generic or targeted intervention). They will receive either targeted ("Countdown: Preparing to Quit Smoking with Low-Nicotine Cigarettes") or generic ("Clearing the Air") materials, and will receive one-on-one counseling.
  Very Low Nicotine Content (VLNC) Cigarettes: Eligible participants will receive a 1-week supply (based on typical # cigarettes/day x 1.5) of normal nicotine content (NNC) (.8 mg nicotine yield) study cigarettes to smoke exclusively during one baseline week.
  Study 1: Participants (n=20) will then be randomly selected to receive either the lowest nicotine dose of VLNC cigarettes, or gradual decreasing nicotine VLNC cigarettes, ten participants per each group, over the next four weeks.
  Study 2: Participants (n=208) will be randomly assigned to 1 of 4 Study 2 Reduction Arms, 52 participants per arm.
  One on One Counseling: All participants will receive One on One Counseling.
Arm/Group | Study 2: Targeted/Immediate Reduction | Study 2: Targeted/Gradual Reduction | Study 2: Generic/Immediate Reduction | Study 2: Generic/Gradual Reduction
Number analyzed (Participants) | 41 | 32 | 34 | 40
participants | 12 | 8 | 10 | 13

3. Primary Outcome: Study 2 - Participant Abstinence Success at 6 Months
Description: Participants reporting 7-day point prevalence abstinence at 6 months
  RCT: The purpose of Study 2 is to test effects of the targeted intervention developed in Study 1 on smoking cessation. Comparison of abstinence success per treatment arm, utilizing 7-day point prevalence abstinence at each follow-up assessment.
Time Frame: At 6 Months
Measure: Number; unit: participants
Arm/Group | Study 2: Targeted/Immediate Reduction | Study 2: Targeted/Gradual Reduction | Study 2: Generic/Immediate Reduction | Study 2: Generic/Gradual Reduction
Number analyzed (Participants) | 41 | 32 | 34 | 40
participants | 10 | 7 | 6 | 10

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from date of on study to when participant has last study visit, approximately 6 months.
Arm/Group | Study 1: Immediate Reduction | Study 1: Gradual Reduction | Study 2: Targeted/Immediate Reduction | Study 2: Targeted/Gradual Reduction | Study 2: Generic/Immediate Reduction | Study 2: Generic/Gradual Reduction
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/41 | 0/32 | 0/34 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/41 | 3/32 | 1/34 | 2/40
Other Adverse Events (participants affected / at risk) | 5/7 | 3/8 | 25/41 | 20/32 | 24/34 | 27/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study 1: Immediate Reduction (N=7) | Study 1: Gradual Reduction (N=8) | Study 2: Targeted/Immediate Reduction (N=41) | Study 2: Targeted/Gradual Reduction (N=32) | Study 2: Generic/Immediate Reduction (N=34) | Study 2: Generic/Gradual Reduction (N=40)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study 1: Immediate Reduction (N=7) | Study 1: Gradual Reduction (N=8) | Study 2: Targeted/Immediate Reduction (N=41) | Study 2: Targeted/Gradual Reduction (N=32) | Study 2: Generic/Immediate Reduction (N=34) | Study 2: Generic/Gradual Reduction (N=40)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 5 (6) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 1 (1) | 0 (0)
Tooth discoloration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 3 (3) | 3 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carbon monoxide diffusing capacity decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 6 (8)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus pain (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 3 (4) | 6 (7)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (6) | 8 (9) | 5 (5) | 7 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (5) | 3 (4) | 5 (6) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 9 (11) | 5 (5) | 5 (8)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urticaria (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell spot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT02796391/Prot_SAP_000.pdf